CLINICAL TRIAL: NCT06804044
Title: Effects of Different Dietary Programs on Anthropometric Parameters in Women With Polycystic Ovary Syndrome
Brief Title: Intermittent Fasting (IF) Has Gained Recognition as a Promising Weight Loss Approach That Improves Body Weight, Insulin Resistance, and Metabolism. While Standard Diets Are Common in PCOS Management, IF May Address the Underlying Causes of Weight Gain and Offer Additional Metabolic Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Yonca Sevim, Assistant Professor, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12309112022
Record Dates: First submitted 2025-01-21; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2022-11

CONDITIONS: Polycystic Ovary Syndrome; Weight Loss; Intermittent Fasting; Medical Nutrition Therapy; Caloric Restriction
Keywords: Diet; PCOS; IF
MeSH Terms: conditions — Polycystic Ovary Syndrome; Weight Loss; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent Fasting Diet Therapy (Experimental): The dietary principles implemented for overweight/obese women with PCOS: targeting a 5% weight loss in line with the recommendations of the Turkish Endocrinology and Metabolism Association, calculating daily calorie requirements using the Harris-Benedict formula, and setting macronutrient distribution ratios to 45-60% carbohydrates, 15-20% protein, and 25-30% fat.
  Interventions: Behavioral: Intermittent Fasting
- Standart Diet Therapy (Experimental): The dietary principles implemented for overweight/obese women with PCOS: targeting a 5% weight loss in line with the recommendations of the Turkish Endocrinology and Metabolism Association, calculating daily calorie requirements using the Harris-Benedict formula, and setting macronutrient distribution ratios to 45-60% carbohydrates, 15-20% protein, and 25-30% fat.
  Interventions: Behavioral: Standart Diet Therapy
- Free of dietary intervention (No Intervention): No dietary intervention was made and the individuals continued their current diet.

INTERVENTIONS:
Behavioral: Intermittent Fasting — A 16:8 intermittent fasting with a daytime eating window model was applied.
  Arms: Intermittent Fasting Diet Therapy
Behavioral: Standart Diet Therapy — Meal plan with 3 main meals and 3 snacks was applied.
  Arms: Standart Diet Therapy

SUMMARY:
The goal of this clinical trial is to learn if dietary interventions works to improve anthropometric measures in women with PCOS. The main questions it aims to answer are:

* Does intermittent fasting (IF) cause loss of body weight, fat and muscle mass?
* Can IF be considered more effective to medical and standart nutrition therapy (SDT)?
* What dietary problems do participants have when having IF diet?

Participants will:

* Follow IF, SDT, or no intervention for 8 weeks.
* Visit the clinic once every 2 weeks for check ups with a total of 5 visits for intervention groups IF and STD, visit at the beginning, second week and at the end for control group
* Keep dietary records

DETAILED DESCRIPTION:
It was conducted in individuals who were diagnosed with PCOS as a result of clinical, biochemical and ultrasonographic medical evaluation by a gynecologist.

ELIGIBILITY:
Inclusion Criteria:

* Voluntariness to participate in the study
* BMI between 25-35 kg/m2
* Women between the ages of 18-45

Exclusion Criteria:

* An endocrine disorder other than polycystic ovary syndrome
* Chronic liver and kidney disease,
* Diabetes,
* Hypertension,
* Hyperuricemia,
* Heart Failure,
* Thyroid disease,
* Pregnant and breastfeeding women,
* Individuals with psychiatric disorders,
* Oncological diseases,
* Women using medication,
* Those with pacemakers and platinum,
* Those with special nutritional needs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Body Weight lose | 8 weeks
  Total body weight (kg)
Body Composition: Fat, Muscle | 8 weeks
  Body Muscle= skeletal muscle mass (kg), regional muscle analysis (right-left arm, trunk, right-left leg) (kg).
  Body Fat= fat mass (kg), regional fat analysis (right-left arm, trunk, right-left leg) (kg).
Body Circumference Measurements | 8 weeks
  Waist Circumference, Hip Circumference, Upper Arm Circumference, Neck Circumference

SECONDARY OUTCOMES:
Body Mass Indeks | 8 weeks
  weight (kg) and height (cm) will be combined to report BMI in kg/m^2
Body Fat Ratio | 8 weeks
  total fat ratio (%)
Body Water | 8 weeks
  Body water (ml)
Dietary Energy Intakes | 8 weeks
  Energy (kcal),
Energy Ratio from Macronutrients | 8 weeks
  Carbohydrate energy %, Protein energy % ,Fat energy %
Dietary Macronutrients Intakes | 8 weeks
  Macronutrients: carbohydrates (g), proteins (g), fats (g)
Dietary Micronutrients Intakes | 8 weeks
  Micronutrents: Vitamin and Mineral intakes will be presented as a percentage (%) of meeting the daily recommended intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahçeşehir University, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No